CLINICAL TRIAL: NCT00829790
Title: A Single-Dose, 2-Period, 2-Treatment, 2-Way Crossover Study of Doxycycline Monohydrate 25 mg as a 5mL Oral Suspension Under Fed Conditions
Brief Title: Doxycycline Monohydrate 25 mg (5mL) Oral Suspension Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20-065-SA
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Doxycycline

ARMS (2):
- 1 (Experimental): Doxycycline Monohydrate
  Interventions: Drug: Doxycycline Monohydrate
- 2 (Active Comparator): Vibramycin Monohydrate®
  Interventions: Drug: Doxycycline Monohydrate

INTERVENTIONS:
Drug: Doxycycline Monohydrate — 25 mg 5mL oral dose
  Arms: 1
Drug: Doxycycline Monohydrate — 25 mg 5 mL dose
  Other Names: Vibramycin Monohydrate®
  Arms: 2

SUMMARY:
The objective of this study was to compare the rate of absorption and the oral bioavailability of a test formulation of doxycycline monohydrate 1 x 25 mg (5mL) oral suspension manufactured by IVAX Pharmaceuticals, Inc. and distributed by TEVA Pharmaceuticals USA to an equivalent oral dose of the commercially available reference product, Vibramycin Monohydrate® manufactured by Pfizer, Inc. Following an overnight fast of at least 10 hours, subjects consumed a standard high-calorie. high-fat breakfast meal. This standard breakfast meal began 30 minutes prior to each dose.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria

All subjects must satisfy the following criteria to be considered for study participation:

* Subject must be male or non-pregnant, non-breast-feeding female
* Subject must be at least 18 years of age
* Subject must have a Body Mass Index (BMI) between 18 and 30 kg/m2, inclusive, and body weight should be at least 50 kg (110 lbs)
* Female Subjects - not surgically sterile or at least two years postmenopausal - must agree to utilize one of the following forms of contraception, if sexually active with a male partner, from screening through completion of the study. Approved forms of contraception are abstinence, double barrier (condom with spermicide, diaphragm with spermicide), intra-uterine device (IUD), or vasectomized partner (6 months minimum since vasectomy).
* Subject must voluntarily consent to participate in this study and provide their written informed consent prior to the start of any study-specific procedures.
* Subject is willing and able to consume the entire high-calorie, high-fat breakfast meal in the designated timeframe required during each study period.
* Subject is willing and able to remain in the study unit for the entire duration of each confinement period and return for any outpatient visits.

Exclusion Criteria

Subjects may be excluded for any of the following:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition which, in the opinion of the Investigator would jeopardize the safety of the subject or the validity of the study results.
* Has a clinically significant abnormal finding on the physical exam, medical history, ECG or clinical laboratory results at screening.
* History or presence of allergic or adverse response to doxycycline monohydrate or related drugs.
* Has been on a significantly abnormal diet during the four weeks preceding the first dose of study medication.
* Has donated blood or plasma within 30 days prior to the first dose of study medication.
* Has participated in another clinical trial within 30 days prior to the first dose of study medication.
* Has used any over-the-counter (OTC) medication, including nutritional supplements, within 7 days prior to the first dose of study medication.
* Has used any prescription medication, including hormonal contraceptive or hormonal replacement therapy, within 14 days prior to the first dose of study medication.
* Has been treated with any known enzyme altering drugs such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication.
* Has smoked or used tobacco products within 90 days prior to the first dose of study medication.
* Is a female with a positive pregnancy test result.
* Has an intolerance to venipuncture.
* Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates)
* Has a history of drug or alcohol abuse.
* Has had a positive test for, or has been treated for hepatitis B, hepatitis C or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-10; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick A Bieberdorf, M.D., Principal Investigator — CEDRA Clinical Research
Locations (1):
- CEDRA Clinical Research, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxycycline Monohydrate First: 25mg(5mL) Doxycycline Monohydrate Oral Suspension test product dosed in first period followed by 25mg(5mL) Vibramycin® Monohydrate Oral Suspension reference product dosed in the second period.
- Vibramycin® Monohydrate First: 25mg(5mL) Vibramycin® Monohydrate Oral Suspension reference product dosed in first period followed by 25mg(5mL) Doxycycline Monohydrate Oral Suspension test product dosed in the second period.
Period: First Intervention
Arm/Group | Doxycycline Monohydrate First | Vibramycin® Monohydrate First
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Washout of 14 Days
Arm/Group | Doxycycline Monohydrate First | Vibramycin® Monohydrate First
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Doxycycline Monohydrate First | Vibramycin® Monohydrate First
Started | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxycycline Monohydrate First | Vibramycin® Monohydrate First | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 5 | 8 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 1 | 3 | 4
  White | 4 | 8 | 12
  Hispanic | 9 | 4 | 13
  More than One | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Cmax = Maximum Observed Concentration.
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Doxycycline Monohydrate: 25mg(5mL) Doxycycline Monohydrate Oral Suspension test product dosed in either period.
- Vibramycin® Monohydrate: 25mg(5mL) Vibramycin® Monohydrate Oral Suspension reference product dosed in either period.
Arm/Group | Doxycycline Monohydrate | Vibramycin® Monohydrate
Number analyzed (Participants) | 29 | 29
ng/mL | 295 (77.8) | 256 (65.5)
Statistical Analysis 1: Comparison: Doxycycline Monohydrate vs Vibramycin® Monohydrate; Test type: Non-Inferiority or Equivalence — The ANOVA model was utilized in comparing the effects between the test and reference products. Differences were declared statistically significant at the 5% level (p<0.05); Ratio of the T/R geometric mean x 100 = 114.49, 90% CI [109.25 to 119.98] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t = Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration.
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Doxycycline Monohydrate | Vibramycin® Monohydrate
Number analyzed (Participants) | 29 | 29
ng*h/mL | 5869 (1449) | 4991 (1216)
Statistical Analysis 1: Comparison: Doxycycline Monohydrate vs Vibramycin® Monohydrate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 117.16, 90% CI [110.44 to 124.28] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf = Area Under the Concentration-time Curve From Time Zero to Infinity.
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Doxycycline Monohydrate | Vibramycin® Monohydrate
Number analyzed (Participants) | 29 | 29
ng*h/mL | 6330 (1417) | 5413 (1206)
Statistical Analysis 1: Comparison: Doxycycline Monohydrate vs Vibramycin® Monohydrate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 116.7, 90% CI [109.89 to 123.92] — [estimate comment as in outcome 1, analysis 1]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.